CLINICAL TRIAL: NCT04782024
Title: A Randomized, Double-Blind, Placebo Controlled Parallel Study to Investigate the Effect of 7-Keto on Resting Metabolic Rate in Overweight Adults
Brief Title: A Study to Investigate the Effect of 7-Keto on Resting Metabolic Rate in Overweight Adults
Acronym: 15KMHI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: InterHealth Nutraceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15KMHI
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Resting Metabolic Rate; Overweight Subjects
Keywords: Resting Metabolic Rate; 7-Keto-DHEA; Efficacy; Overweight Adults; Obese Adults

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- 7-Keto 50mg (Experimental)
  Interventions: Dietary Supplement: 7-Keto 50mg
- 7-Keto 25mg (Experimental)
  Interventions: Dietary Supplement: 7-Keto 25mg

INTERVENTIONS:
Dietary Supplement: 7-Keto 50mg
  Arms: 7-Keto 50mg
Dietary Supplement: 7-Keto 25mg
  Arms: 7-Keto 25mg
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the effect of two different doses of 7-Keto compared to placebo on resting metabolic rate. One third of subjects will be given the lower 7-Keto dose, one third will be given the higher 7-Keto dose and one third will be given the placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 20 to 55 years of age
2. If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

   OR

   Female subject of childbearing potential must agree to use a medically approved method of non-hormonal birth control and have a negative urine pregnancy test result. Birth Control methods must be initiated at least 14 days prior to randomization and must be continued until 28 days after the end of study visit. Acceptable methods of birth control include:
   * Double barrier method
   * Intrauterine devices (non-hormonal)
   * Cervical caps or sponges
   * Use of male/female condom
   * Vasectomy of partner
   * Non-heterosexual lifestyle
3. If female and currently experiencing menstrual cycles, subjects should have regular menstrual cycles (28 ± 2 days) and must be in their follicular phase during the duration of the study period (i.e. baseline to visit 3)
4. BMI 25-34.9 ±1 kg/m2
5. Stable weight defined as less than 5kg (approx. 11lbs) gained or lost in the past 3 months
6. Sedentary subjects; defined as subjects with a desk/inactive job, not engaging in any regular sports or exercise programs either at an exercise facility or at home. Occasional activity, low intensity yoga and walking at a regular pace are acceptable.
7. Agreement to maintain current level of physical activity through the study and avoid exercising 24 hours prior to study visits
8. Agreement to adopt a diet with a 500 kcal reduction for the duration of the study period.
9. Agreement to completely avoid caffeine consumption, such as coffee, tea and soft drinks 24 hours before study visits and to limit consumption of coffee, tea and soft drinks to 2 cups per day for all other days during the study.
10. Agreement to completely avoid consumption of energy drinks for 24 hours before the screening and baseline visits and for the duration of the study.
11. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Immunodeficiency (i.e. HIV positive, rheumatoid arthritis, history of organ transplant)
3. Use of tobacco products and nicotine products.
4. Use of prescription, over-the-counter, or natural health products known to affect weight and/or metabolic rate within 4 weeks of randomization and during the trial
5. Unstable medical conditions
6. Uncontrolled blood pressure (i.e. systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg)
7. Type I or II diabetes, metabolic disease or any condition that in the opinion of the Qualified Investigator does not safely allow for a reduction in calorie intake
8. Any evidence of an eating disorder, such as anorexia or bulimia, or the presence of any illness that might represent a potential cause of weight loss
9. Abnormal ECG at screening
10. Clinically significant abnormal laboratory results at screening (e.g. AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN; serum creatinine > 1.5 x ULN)
11. Currently taking anti-psychotic medication
12. Participation in a clinical research trial within 30 days prior to randomization
13. Allergy or sensitivity to study supplement ingredients
14. Alcohol abuse (>2 standard alcoholic drinks per day)
15. Current drug abuse or drug abuse within the past 6 months
16. Use of marijuana for medical purposes
17. Individuals who are cognitively impaired and/or who are unable to give informed consent
18. Any other condition, which in the Investigator's opinion, may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Change in resting metabolic rate | 1 week: from baseline to end of study

SECONDARY OUTCOMES:
Change in total body water | 1 week: from baseline to end of study
Change in total body fat | 1 week: from baseline to end of study

OTHER OUTCOMES:
Number of incidents of abnormal lab results | 1 week: from baseline to end of study
  Lab results from blood biochemistry and hematology (Na, K, Cl, creatinine, BUN, AST, ALT, GGT and bilirubin)
Number of incidents of adverse events | 1 week: from baseline to end of study
Change in BMI | 1 week: from baseline to end of study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - KGK USA, Foothill Ranch, California
  - KGK USA, Orlando, Florida